CLINICAL TRIAL: NCT05167526
Title: A Phase 1 Combined Single and Multiple Ascending Oral Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of ASP8731 in Healthy Adult Participants, Including an Assessment of a Food Effect
Brief Title: A Study to Find a Suitable Dose of ASP8731 and Check for Medical Problems at Each Dose in Healthy Adults
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The study was terminated due to protocol defined stopping criteria being met.
Sponsor: Astellas Pharma Global Development, Inc. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Basic Science
Other Study IDs: 8731-CL-0101
Record Dates: First submitted 2021-12-20; First posted 2021-12-22 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Healthy Participants
Keywords: Healthy Participants; Pharmacokinetics; Pharmacodynamics

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Part 1: ASP8731 Placebo (Placebo Comparator): Participants receive a single dose of matching placebo under fasting conditions.
  Interventions: Drug: ASP8731 Matching Placebo
- Part 1: ASP8731 3mg (Experimental): Participants receive a single dose of ASP8731 3mg under fasting conditions.
  Interventions: Drug: ASP8731
- Part 1: ASP8731 12mg (Experimental): Participants receive a single dose of ASP8731 12 mg under fasting conditions.
  Interventions: Drug: ASP8731
- Part 2: Placebo (Placebo Comparator): Participants receive a multiple matching dose of placebo twice daily for 14 days under fasting conditions.
  Interventions: Drug: ASP8731 Matching Placebo
- Part 2: ASP8731 6mg (Experimental): Participants receive ASP8731 6mg twice daily for 14 days under fasting conditions.
  Interventions: Drug: ASP8731
- Part 1: ASP8731 6mg (Experimental): Participants receive a single dose of ASP8731 6 mg of under fasting conditions.
  Interventions: Drug: ASP8731

INTERVENTIONS:
Drug: ASP8731 — Oral
  Arms: Part 1: ASP8731 12mg; Part 1: ASP8731 3mg; Part 1: ASP8731 6mg; Part 2: ASP8731 6mg
Drug: ASP8731 Matching Placebo — Oral
  Arms: Part 1: ASP8731 Placebo; Part 2: Placebo

SUMMARY:
ASP8731 is a potential new treatment for people with sickle cell disease. Before ASP8731 is available as a treatment, the researchers need to understand how it is processed by and acts upon the body. They do this to find a suitable dose and to check for potential medical problems from the treatment. This type of study usually includes healthy adults but can include people with the relevant condition.

The main aim of this study is to learn if healthy adults have any medical problems after taking different doses of ASP8731.

This study will be in 2 parts.

In Part 1, different small groups of people will take lower to higher doses of ASP8731 or a placebo. In this study a placebo looks like ASP8731 but will not have any medicine in it. This is done to find suitable doses of ASP8731 and work out how often it should be taken. Some of this information will be used in Part 2 of the study. The first group will take the lowest dose of ASP8731 or the placebo. A medical expert panel will check the results from this group and decide which ASP8731 dose the next group can take. The panel will do this for each group until all groups have taken ASP8731 or until a suitable dose of ASP8731 has been reached.

In Part 1, people will visit the study clinic 4 times. The first visit is to check if they can take part. People will be asked about their medical history, have a physical exam, and their vital signs checked (pulse rate, temperature, and blood pressure). Also, they will have an ECG to check their heart rhythm and have some blood samples taken for laboratory tests. For women this will include a pregnancy test.

At the second visit, people will stay in the study clinic for a few days. In most groups, people will be picked to take either ASP8731 or the placebo by chance alone. They will fast before taking ASP8731 or the placebo. 1 group will take ASP8731 with food. No-one in that group will take the placebo. After taking ASP8731 or the placebo (or just ASP8731 with food), people in all groups will give blood and urine samples during the next 3 days. Also, they will be checked for any medical problems during their clinic stay.

People will return to the study clinic for a 2 follow-up visits - at about 8 and 30 days after they last took ASP8731 or the placebo. At these visits people will be asked if they have any medical problems. They will have a physical exam, have their vital signs checked (pulse rate, temperature, and blood pressure), and have some blood samples taken for laboratory tests. For women, this will include another pregnancy test.

In Part 2, other different small groups of people will take lower to higher doses of ASP8731 or a placebo. How often it is taken will be worked out from Part 1.The first group will take the lowest dose of ASP8731 or the placebo each day over several days. A medical expert panel will check the results from this group and decide which ASP8731 dose the next group can take. The panel will do this for each group until all groups have taken ASP8731.

In Part 2, people will visit the study clinic 5 times. The first visit is to check if they can take part. People will be asked about their medical history, have a physical exam, and their vital signs checked. Also, they will have an ECG and have some blood samples taken for laboratory tests. For women this will include a pregnancy test.

At the second visit, people will stay in the study clinic for several days. In all groups, people will be picked to take either ASP8731 or the placebo by chance alone. After taking ASP8731 or the placebo, people in all groups will give blood samples throughout their stay. They will give urine samples during the last few days of their stay. Also, they will be checked for any medical problems during their clinic stay. After discharge, people will return to the clinic 4 days later for a third visit. At this visit, they will have some blood samples taken for laboratory tests. Also, they will have their vital signs checked and will be asked if they have any medical problems.

People will return to the study clinic for a 2 follow-up visits - at about 15 and 30 days after they last took ASP8731 or the placebo. At these visits people will be asked if they have any medical problems. They will have a physical exam and have their vital signs checked. They will also have an ECG and have some blood samples taken for laboratory tests. For women, this will include another pregnancy test.

No other visits are planned during this study.

ELIGIBILITY:
Inclusion Criteria:

* Participant has a body mass index (BMI) range of 18.5 to 32.0 kg/m^2, inclusive and weighs at least 50 kg at screening.
* Female participant is not pregnant and at least 1 of the following conditions apply:

  * Not a woman of childbearing potential (WOCBP)
  * WOCBP who agrees to follow the contraceptive guidance from the time of informed consent through at least 30 days after final IP administration.
* Female participant must agree not to breastfeed starting at 90 days prior to screening and throughout the study period and for 30 days after final investigational product (IP) administration.
* Female participant must not donate ova starting at first dose of IP and throughout the study period and for 30 days after final IP administration.
* Male participant with female partner(s) of childbearing potential (including breastfeeding partner[s]) must agree to use contraception throughout the treatment period and for 90 days after final IP administration.
* Male participant must not donate sperm during the treatment period and for 90 days after final IP administration.
* Male participant with pregnant partner(s) must agree to remain abstinent or use a condom for the duration of the pregnancy throughout the study period and for 30 days after final IP administration.
* Participant agrees not to participate in another interventional study while receiving study treatment in the present study.

Exclusion Criteria:

* Participant has received any investigational therapy within 28 days or 5 half lives, whichever is longer, prior to screening.
* Participant has any condition which makes the participant unsuitable for study participation.
* Participant has a known or suspected hypersensitivity to ASP8731 or any components of the formulation used.
* Female participant who has been pregnant within 6 months prior to screening or breastfeeding within 90 days prior to screening.
* Participant has had previous exposure with ASP8731.
* Participant has any of the liver function tests (alkaline phosphatase, alanine aminotransferase, aspartate aminotransferase and total bilirubin) above the upper limit of normal (ULN) on day -1. In such a case, the assessment may be repeated once.
* Participant has any history of previously diagnosed Gilbert's syndrome.
* Participant has creatinine level outside normal limits on day -1. In such a case, the assessment may be repeated once.
* Participant has any clinically significant history of allergic conditions (including drug allergies, asthma, eczema or anaphylactic reactions, but excluding untreated, asymptomatic, seasonal allergies) prior to first IP administration.
* Participant has any history or evidence of any clinically significant cardiovascular, gastrointestinal, endocrinologic, hematologic (e.g., sickle cell disease, hemoglobinopathies, hemolytic anemias, etc.), hepatic, immunologic, metabolic, urologic, pulmonary, neurologic, dermatologic, psychiatric, renal and/or other major disease or malignancy.
* Participant has/had febrile illness or symptomatic, viral, bacterial (including upper respiratory infection) or fungal (noncutaneous) infection within 1 week prior to day -1.
* Participant has any clinically significant abnormality of the physical examination, ECG and protocol-defined clinical laboratory tests at screening or on day -1.
* Participant has a mean pulse < 45 or > 90 bpm; mean systolic blood pressure > 140 mmHg; mean diastolic blood pressure > 90 mmHg (measurements taken in triplicate after participant has been resting in the supine position for at least 5 minutes; pulse will be measured automatically) on day -1. If the mean blood pressure or pulse exceeds the limits above, 1 additional triplicate may be taken.
* Participant has a mean QT corrected for heart rate by Fridericia's cube root formula (QTcF) of > 430 msec (for male participants) and > 450 msec (for female participants) on day -1. If the mean QTcF exceeds the limits above, 1 additional triplicate ECG may be taken.
* Participant has an abnormal heart rhythm such as prolonged QT interval, underlying heart disease, chronic kidney disease or receiving medicines which prolong the QT interval.
* Participant has used any prescribed or nonprescribed drugs (including vitamins, natural and herbal remedies, e.g., St. John's Wort) in the 2 weeks prior to first IP administration, except for occasional use of acetaminophen (up to 2 g/day), topical dermatological products (including corticosteroid products), hormonal contraceptives and hormone replacement therapy (HRT).
* Participant has smoked, used tobacco-containing products or nicotine containing products (e.g., electronic vapes) within 6 months prior to screening or the participant tests positive for cotinine at screening or on day -1.
* Participant has a history of consuming > 14 units for male participants or > 7 units for female participants of alcoholic beverages per week within 6 months prior to screening or has a history of alcoholism or drug/chemical/substance abuse within 2 years prior to screening (note: 1 unit = 12 ounces of beer, 4 ounces of wine, 1 ounce of spirits/hard liquor) or the participant tests positive for alcohol at screening or on day -1.
* Participant has used any drugs of abuse (amphetamines, barbiturates, benzodiazepines, cannabinoids, cocaine and/or opiates) within 3 months prior to day -1 or the participant tests positive for drugs of abuse (amphetamines, barbiturates, benzodiazepines, cannabinoids, cocaine and opiates) at screening or on day -1.
* Participant has consumed more than 400 mg of caffeine (4 cups of coffee) per day in the 48 hours prior to first IP administration on day 1 and/or is unwilling to abstain from coffee (or caffeine-containing product) consumption through discharge from unit.
* Participant has used any inducer of metabolism (e.g., barbiturates and rifampin) in the 3 months prior to day -1.
* Participant has had significant blood loss, donated ≥ 1 unit (450 mL) of whole blood or donated plasma within 7 days prior to day -1 and/or received a transfusion of any blood or blood product within 60 days.
* Participant has a positive serology test for hepatitis A virus (HAV) antibodies (IgM), hepatitis B core (HBc) antibodies, hepatitis B surface antigen (HBsAg), hepatitis C virus (HCV) antibodies or antibodies to human immunodeficiency virus (HIV) type 1 and/or type 2 at screening.
* Participant has received a coronavirus disease 2019 (COVID-19) vaccine within the 2 weeks prior to first IP administration or will have a COVID-19 vaccine dose before the follow-up visit 2.
* Participant has a positive result for severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) polymerase chain reaction (PCR) test at screening or on day 1.
* Participant is an employee of Astellas, the study-related contract research organizations (CROs) or the clinical unit.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2022-03-07 (Actual); Primary Completion 2022-11-10 (Actual); Study Completion 2022-11-10 (Actual)

PRIMARY OUTCOMES:
Part 1: Safety and tolerability assessed by nature, frequency, and severity of Adverse Events (AEs) | Up to Day 41
  Adverse Events (AEs) will be coded using medical dictionary for regulatory activities (MedDRA). An AE is any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of study IP, whether or not considered related to the study investigational product (IP). An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of study IP. This includes events related to the comparator and events related to the (study) procedures.
Part 1: Number of participants with laboratory value abnormalities and/or adverse events (AEs) | Up to Day 41
  Number of participants with potentially clinically significant laboratory values.
Part 1: Number of participants with vital sign abnormalities and/or adverse events (AEs) | Up to Day 41
  Number of participants with potentially clinically significant vital sign values.
Part 1: Number of participants with electrocardiogram (ECG) abnormalities and/or adverse events | Up to Day 41
  Number of participants with potentially clinically significant ECG values.
Part 2: Safety and tolerability assessed by nature, frequency, and severity of Adverse Events (AEs) | Up to Day 59
  Adverse Events (AEs) will be coded using medical dictionary for regulatory activities (MedDRA). An AE is any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of study IP, whether or not considered related to the study investigational product (IP). An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of study IP. This includes events related to the comparator and events related to the (study) procedures.
Part 2: Number of participants with laboratory value abnormalities and/or adverse events (AEs) | Up to Day 59
  Number of participants with potentially clinically significant laboratory values.
Part 2: Number of participants with vital sign abnormalities and/or adverse events (AEs) | Up to Day 59
  Number of participants with potentially clinically significant vital sign values.
Part 2: Number of participants with electrocardiogram (ECG) abnormalities and/or adverse events | Up to Day 59
  Number of participants with potentially clinically significant ECG values.

SECONDARY OUTCOMES:
Part 1: Pharmacokinetics (PK) of ASP8731 in plasma: area under the concentration-time curve from the time of dosing extrapolated to time infinity (AUCinf) | Up to Day 7
  AUCinf will be recorded from the PK plasma sample collected.
Part 1: PK of ASP8731 in plasma: area under the concentration-time curve from the time of dosing to the last measurable concentration (AUClast) | Up to Day 7
  AUClast will be recording from the PK plasma sample collected.
Part 1: PK of ASP8731 in plasma: maximum concentration (Cmax) | Up to Day 7
  Cmax will be recorded from the PK plasma sample collected.
Part 2: First Dose PK of ASP8731 in plasma: area under the concentration-time curve from the time of dosing to 24 hours (AUC24) | Up to Day 2
  AUC24 will be recorded from the PK plasma sample collected.
Part 2: First Dose PK of ASP8731 in plasma: area under the concentration-time curve from the time of dosing to 12 hours (AUC12) | Up to Day 2
  AUC12 will be recorded from the PK plasma sample collected.
Part 2: First Dose PK of ASP8731 in plasma: maximum concentration (Cmax) | Up to Day 2
  Cmax will be recorded from the PK plasma sample collected.
Part 2: Last Dose PK of ASP8731 in plasma: area under the concentration-time curve during a dosing interval, where tau (t) is the length of the dosing interval (AUCtau) | Up to Day 20
  AUCtau will be recorded from the PK plasma sample collected.
Part 2: Last Dose PK of ASP8731 in plasma: maximum concentration (Cmax) | Up to Day 20
  Cmax will be recorded from the PK plasma sample collected.
Part 2: Last Dose PK of ASP8731 in plasma: concentration immediately prior to dosing at multiple dosing (Ctrough) | Up to Day 20
  Ctrough will be recorded from the PK plasma sample collected.
Part 2: Morning Dose PK of ASP8731: concentration immediately prior to dosing at multiple dosing (Ctrough) | Up to Day 14
  Ctrough will be recorded from the PK sample collected.
Part 2: Evening Dose PK of ASP8731: concentration immediately prior to dosing at multiple dosing (Ctrough) | Up to Day 12
  Ctrough will be recorded from the PK sample collected.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director Medical Specialties, Study Director — Astellas Pharma Global Development, Inc.
Locations (1):
- California Clinical Trials Medical Group, Glendale, California, United States

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.